CLINICAL TRIAL: NCT04581135
Title: Prospective Observational Cohort Study to Investigate Long-term Pulmonary and Extrapulmonary Effects of COVID-19
Brief Title: Study to Investigate Long-term Pulmonary and Extrapulmonary Effects of COVID-19
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00799
Record Dates: First submitted 2020-09-17; First posted 2020-10-09 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
Keywords: COVID-19; Coronavirus infection; Lung abnormalities; Radiological abnormalities; ARDS; Quality of Life
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples Without DNA — Coded biological material
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 Lung: COVID-19 survivors in Switzerland
  Interventions: Other: COVID-19

INTERVENTIONS:
Other: COVID-19 — Research project in which biological material is sampled and health-related personal data are collected and used for further research. Coded data are used.
  Other Names: Sampling biological material; Collection of health-related personal data

SUMMARY:
Prospective Observational Swiss Cohort Study to Investigate Long-term Pulmonary and Extrapulmonary Effects of COVID-19.

DETAILED DESCRIPTION:
COVID-19 is a coronavirus induced viral pneumonia leading to Acute Respiratory Distress Syndrome. Previous coronavirus infections (SARS and MERS) led to pulmonary fibrosis in up to 30%. Prospective evaluation of lung abnormalities and pulmonary fibrosis after COVID-19 infection is crucial as novel treatments against lung fibrosis of different etiologies are available. No data on pulmonary longterm effects in COVID-19 survivors are currently available. The nation-wide Swiss COVID-19 lung group establishes a meticulously characterized prospective cohort study on pulmonary long-term sequela of patients living in Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* All adult patients with COVID-19 over 18 years.

Exclusion Criteria:

* Severe mental or physical disability precluding informed consent or compliance with the protocol for prospective data collection.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included are survivors of COVID-19.
Sampling Method: Probability Sample
Enrollment: 620 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Pulmonary follow-up sequelae in patients after COVID-19 | 36 months
  Number of patients with the long-term pulmonary complications by measuring lung function, exercise testing and radiological Imaging
Evaluation of risk factors for adverse Outcome after COVID-19 | 36 months
  Number of patients with risk factors including comorbidities and other cofactors and correlate them to adverse outcome in patients after COVID-19

SECONDARY OUTCOMES:
Compare the functional Pulmonary outcome of COVID-19 disease | 36 months
  Compare pulmonary function measurements between mild and moderate to severe and critical COVID-19 disease
Compare the radiological Pulmonary outcome of COVID-19 disease | 36 months
  Compare imaging measurements between mild and moderate to severe and critical COVID-19 disease
Quality of Life after COVID-19 | 36 months
  Compare Quality of Life questionnaires between mild and moderate to severe and critical COVID-19 disease
Physical performance after COVID-19 using Clinical Frailty Scale | 36 months
  To observe and compare the physical performance after COVID-19 via the Clinical Frailty Scale between mild and moderate to severe and critical COVID-19 disease
Physical performance after COVID-19 using frailty assessment tests | 36 months
  To observe and compare the physical performance after COVID-19 via frailty assessment tests between mild and moderate to severe and critical COVID-19 disease
Microbiota and COVID-19 | 36 months
  Number of patients with changes in microbiota in response to COVID-19 by microbiota analysis of sputa, bronchoalveolar lavage and swaps

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Funke-Chambour, MD, Principal Investigator — University Hospital Bern, Department of Pulmonary Medicine - Lead Center
Locations (9):
- Switzerland (9):
  - St. Claraspital AG - Department of Pulmonary Medicine, Basel
  - Universtiy Hospital Bern (Inselspital), Department of Pulmonary Medicine - Lead Center, Bern
  - University and Hospital of Fribourg, Fribourg
  - Hôpitaux Universitaires de Genève - Service de Pneumologie, Geneva
  - CHUV - Service de Pneumologie, Lausanne
  - Clinica Moncucco, Lugano
  - Kantonspital St. Gallen - Klinik für Pneumologie und Schlafmedizin Lungenzentrum, Sankt Gallen
  - Hôpital du Valais - Service de Pneumologie, Sion
  - Universitätsspital Zürich - Klinik für Pneumologie, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abu Hussein N, Machahua C, Ruchti SC, Horn MP, Piquilloud L, Prella M, Geiser TK, von Garnier C, Funke-Chambour M. Circulating calprotectin levels four months after severe and non-severe COVID-19. BMC Infect Dis. 2023 Oct 3;23(1):650. doi: 10.1186/s12879-023-08653-7. PMID 37789266